CLINICAL TRIAL: NCT02847793
Title: Changes in Selective Attentional Patterns Towards Emotional Stimuli by Using Eye-tracking Techniques: A New Intervention for Depression
Brief Title: Attentional Bias Modification Through Eye-tracker Methodology (ABMET)
Acronym: ABMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Carmelo Vázquez, Full Professor of Psychopathology, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PSI2014-61764-EXPLORA
Record Dates: First submitted 2016-07-22; First posted 2016-07-28 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Cognitive Deficits; Depression; Alteration of Cognitive Function
Keywords: Attentional Bias Modification (ABM); Cognitive Bias Modification (CBM); Depression; Dysphoria; Gaze patterns; Eye-tracking
MeSH Terms: conditions — Cognition Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gaze training (Active Comparator): Participants are required to maintain their gaze in a given picture (e.g., a happy face), for a given time (i.e., 750ms vs 1500 ms) to advance to the next trial
  Interventions: Behavioral: Gaze training
- Placebo intervention (Placebo Comparator): Using a matching procedure (i.e., yoked control group), participants are required to maintain their gaze in a given picture (e.g., a happy face), for the same average time that their counterparts in the Gaze training group (i.e. Experimental group)
  Interventions: Behavioral: Placebo intervention

INTERVENTIONS:
Behavioral: Gaze training — Participants are required to maintain their gaze in a given picture (e.g., a happy face), for a given time (i.e., 750ms vs 1500 ms) to advance to the next trial. (A total of 576 trials will be distributed in a 2-day intervention).
  Other Names: Attentional Bias Modification (ABM)
  Arms: Gaze training
Behavioral: Placebo intervention — Participants are exposed to the same amount of time to the experimental stimuli used in the experimental group but there is no contingency between participants' gaze patterns and the end of each of the 576 trials.
  Arms: Placebo intervention

SUMMARY:
Cognitive biases are a hallmark of depression but there is scarce research on whether these biases can be directly modified by using specific cognitive training techniques.

The aim of this study will be targeting and modifying specifically relevant attention biases in participants with subclinical depression using eye-tracking methodologies. This innovative approach has been proposed as a promising future line of intervention in Attention Bias Modification procedures (Koster & Hoorelbeke, 2015).

Recent findings suggest that depression is characterized by a double attentional bias (Duque & Vazquez, 2015), More specifically, depressed individuals have difficulties both to disengage from negative materials (e.g., sad faces) and to engage with positive materials (e.g., happy faces). Thus, training procedures to change attentional biases should target these two separate components.

DETAILED DESCRIPTION:
The aim of this study will be to apply eye-tracking methods to modify specific components of attentional bias in depression. Eye-tracking technology enables us to train attention by following strict performance and time-based criteria as well as to specify the components of attention (i.e., disengagement from negative information, engagement and maintenance in positive information) to be targeted in the training, critical to providing a theory-driven intervention (Koster, Baert et al., 2010). In the case of depression, there is also some evidence from eye-tracking studies showing that recovery from an induced negative mood is better when individuals spontaneously direct their gaze towards positive stimuli (Sanchez et al., 2014). Thus extant evidence on attentional biases in depression suggest that modification of these biases could be a fruitful way to change participants' mood.

Although initial positive results of ABM led some authors to propose it as an alternative treatment for emotional disorders (Bar-Haim, 2010; MacLeod & Holmes, 2012), some recent meta-analysis (Mogoase et al. 2014; Cristea et al., 2015) have reduced the enthusiasm of those previous claims.Yet, it is likely that modest results of ABM procedures in depression are, in part, based on flawed methodologies. The proposed study aims to rectify several limitations of previous designs while opening a new strategy, based in training ocular movements, to modify attentional patterns. With a series of methodological and conceptual improvements (i.e., trial-by- trial feedback, use of different tasks to measure attentional bias and to do the ABM, use of a yoked-group design to control for the time exposure to the emotional stimuli in the control group, and use of a stress-test to measure transfer of the training to a different task), it is expected that some limitations found in previous studies can be overcome. The general aim of the study will be to train adaptive attentional biases (i.e., training the maintenance of gaze towards positive stimuli). The use of the new ABM in a sample of dysphoric participants will allow us to test if training visual selective attention using eye-tracking methodology could be a promising venue for future ABM procedures more solidly grounded on current theories of depression.

ELIGIBILITY:
Inclusion Criteria:

* A score of >13 in the Beck Depression Inventory (BDI-II)

Exclusion Criteria:

* Impaired vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Assessment of current mood (PANAS) | Change from Baseline to the end of the 2-day intervention.It will be administered 12 min before the first session of training and then immediately after finishing the 2nd session of training
  A scale measuring current general positive and negative mood
Assessment of current mood (EVEA) | Change from Baseline to the end of the 2-day intervention. It will be administered 12 min before the first session of training and then immediately after finishing the 2nd session of training.
  A scale measuring current anger, happiness, anxiety and depressed mood
Attentional Bias Assessment Task (ABA, Sanchez et al., 2013) | Change from Baseline to the end of the 2-day intervention. It will be administered immediately before the first session of training and then 5 min after finishing the 2nd session of training
  An eye-tracking task to measure gaze patterns towards emotional faces

SECONDARY OUTCOMES:
Beck Depression Inventory-II | Change from Baseline to the end of the 2-day intervention. It will be administered 20 min before the first session of training and then 20 min after finishing the 2nd session of training
  Symptoms of depression
Beck Anxiety Inventory | Change from Baseline to the end of the 2-day intervention. It will be administered 20 min before the first session of training and then 20 min after finishing the 2nd session of training.
  Symptoms of anxiety
Ruminative Responses Scale (RRS) | Change from Baseline to the end of the 2-day intervention. It will be administered 20 min before the first session of training and then 20 min after finishing the 2nd session of training
  Ruminative style
White Bear Suppression Inventory (WBSI) | Change from Baseline to the end of the 2-day intervention. It will be administered 20 min before the first session of training and then 20 min after finishing the 2nd session of training.
  Tendency to suppress distressing thoughts and images
Behavioral Activation System (BAS)- Behavioral Inhibition System (BIS) Scale | Change from Baseline to the end of the 2-day intervention. It will be administered 20 min before the first session of training and then 20 min after finishing the 2nd session of training.
  A single scale measuring attitudes and behaviors related to the Behavioral Activation System and the Behavioral Items related to sensitivity to punishment and rewards
Pemberton Happiness Index | Change from Baseline to the end of the 2-day intervention. It will be administered 20 min before the first session of training and then 20 min after finishing the 2nd session of training.
  Integrative measure of well-being
Satisfaction with Life Scale (SWLS) | Change from Baseline to the end of the 2-day intervention. It will be administered 20 min before the first session of training and then 20 min after finishing the 2nd session of training.
  Life satisfaction
Life Orientation Test-Revised (LOT-R) | Change from Baseline to the end of the 2-day intervention. It will be administered 20 min before the first session of training and then 20 min after finishing the 2nd session of training.
  Dispositional optimism

OTHER OUTCOMES:
Emotional Threshold Detection Task (ETDT). | Change from Baseline to the end of the 2-day intervention. It will be administered 15 min before the first session of training and then 15 min after finishing the 2nd session of training
  A morphing task to assess changes in participants' participants' thresholds to detect changes in the facial expression of emotions.
Anagram Stress Task (AST) | Immediately after the intervention (i.e., after finishing the 2nd session of training). It will be administered 30 min after finishing the 2nd session of training
  Behavioral persistence in trying to solve anagrams with different levels of difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Vazquez, Ph.D:, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- School of Psychology, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cristea IA, Kok RN, Cuijpers P. Efficacy of cognitive bias modification interventions in anxiety and depression: meta-analysis. Br J Psychiatry. 2015 Jan;206(1):7-16. doi: 10.1192/bjp.bp.114.146761. PMID 25561486
- [Background] Mogoase C, David D, Koster EH. Clinical efficacy of attentional bias modification procedures: an updated meta-analysis. J Clin Psychol. 2014 Dec;70(12):1133-57. doi: 10.1002/jclp.22081. Epub 2014 Mar 20. PMID 24652823
- [Background] Emmelkamp PM. Attention bias modification: the Emperor's new suit? BMC Med. 2012 Jun 25;10:63. doi: 10.1186/1741-7015-10-63. PMID 22731990
- [Background] Macleod C, Holmes EA. Cognitive bias modification: an intervention approach worth attending to. Am J Psychiatry. 2012 Feb;169(2):118-20. doi: 10.1176/appi.ajp.2011.11111682. No abstract available. PMID 22318791
- [Background] Duque A, Vazquez C. Double attention bias for positive and negative emotional faces in clinical depression: evidence from an eye-tracking study. J Behav Ther Exp Psychiatry. 2015 Mar;46:107-14. doi: 10.1016/j.jbtep.2014.09.005. Epub 2014 Sep 22. PMID 25305417
- [Background] Sanchez A, Vazquez C, Marker C, LeMoult J, Joormann J. Attentional disengagement predicts stress recovery in depression: an eye-tracking study. J Abnorm Psychol. 2013 May;122(2):303-13. doi: 10.1037/a0031529. Epub 2013 Feb 18. PMID 23421524
- [Background] Bar-Haim Y, Holoshitz Y, Eldar S, Frenkel TI, Muller D, Charney DS, Pine DS, Fox NA, Wald I. Life-threatening danger and suppression of attention bias to threat. Am J Psychiatry. 2010 Jun;167(6):694-8. doi: 10.1176/appi.ajp.2009.09070956. Epub 2010 Apr 15. PMID 20395400
- [Derived] Vazquez C, Blanco I, Sanchez A, McNally RJ. Attentional bias modification in depression through gaze contingencies and regulatory control using a new eye-tracking intervention paradigm: study protocol for a placebo-controlled trial. BMC Psychiatry. 2016 Dec 8;16(1):439. doi: 10.1186/s12888-016-1150-9. PMID 27931196